CLINICAL TRIAL: NCT03895853
Title: Early Metabolic Resuscitation: A Potential Solution to Multi-Organ Dysfunction Syndrome in Septic Shock
Brief Title: Early Metabolic Resuscitation for Septic Shock
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: At the request of the PI
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0986; NCI-2019-01392 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0986 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2021-03

CONDITIONS: Multiple Organ Failure; Septic Shock; Severe Sepsis
MeSH Terms: conditions — Multiple Organ Failure; Shock, Septic; Sepsis | interventions — Practice Guidelines as Topic; Standard of Care; Parenteral Nutrition; Glucose; Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (standard of care) (Active Comparator): Patients receive standard of care for septic shock.
  Interventions: Other: Best Practice
- Group II (early metabolic resuscitation) (Experimental): Patients receive standard of care treatment for septic shock and early metabolic resuscitation (IV) over continuous infusion for up to 7 days.
  Interventions: Other: Best Practice; Dietary Supplement: early metabolic resuscitation

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Dietary Supplement: early metabolic resuscitation — Given Intravenous
  Other Names: hyperalimentation; EMR; glucose; protein; essential metabolic molecules
  Arms: Group II (early metabolic resuscitation)

SUMMARY:
This phase II trial studies how well early metabolic resuscitation therapy works in reducing multi-organ dysfunction in patients with septic shock. Early metabolic resuscitation is made of large doses of glucose, protein, and essential metabolic molecules that may help lower the effects of septic shock on the body. Giving patients early metabolic resuscitation in combination with standard of care may work better in reducing multi-organ dysfunction syndrome in patients with septic shock compared to standard of care alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of administering early metabolic resuscitation with standard of care (SC + EMR) in patients diagnosed with septic shock for reducing 28-day mortality versus using the standard of care alone (SC).

SECONDARY OBJECTIVES:

I. To assess whether early metabolic resuscitation with standard of care (SC + EMR) is an effective strategy to reduce intensive care unit (ICU) mortality, hospital mortality, and 90-day mortality of septic shock patients relative to SC.

II. To compare the time to death from any cause between patients administered SC + EMR versus SC after being diagnosed with septic shock.

III. To assess whether SC + EMR is an effective strategy to reduce complications of septic shock such as: i) acute kidney injury, ii) dialysis requirements, iii) need for cardiovascular support or days on vasopressors, iv) need for invasive ventilation, days on ventilator support, v) duration of ICU stay, and vi) duration of hospital stay versus SC.

IV. To describe the presence of any adverse effects between the two study groups (SC + EMR group versus [vs] SC group); thus, characterizing their safety.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive standard of care for septic shock.

GROUP II: Patients receive standard of care treatment for septic shock and early metabolic resuscitation (IV) over continuous infusion for up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the adult medical intensive care unit (MICU).
* Diagnosis of septic shock within 12 hours of ICU admission defined as meeting criteria for sepsis in addition to the following: A) Vasopressor therapy needed to elevate mean arterial pressure (MAP) >= 65 mmg Hg. B) Lactate > 2 mmol/L (18 mg/dL) after adequate fluid resuscitation.
* Sequential Organ Failure Assessment (SOFA) score meeting the following requirements A) Cardiovascular SOFA >= 2 B) Total SOFA score =< 12.
* Patients meeting the above and not able to tolerate enteral nutrition above 70% of their estimated daily caloric need.

Exclusion Criteria:

* Do not resuscitate (DNR).
* Comfort care and end-of-life patients.
* Patients with SOFA scores greater than 12.
* Pregnant women.
* Jehovah Witnesses that do not accept albumin.
* Active bleeding (e.g., gastrointestinal bleeding).
* Acute neurological syndromes (e.g., stroke, hemorrhage, etc.).
* End-stage renal disease (ESRD).
* Chronic liver disease

  * Child-Pugh class C
  * Diagnosis of cirrhosis
* Heart rate less than 50 beats per minute (bpm).
* Respiratory rate less than 8 respirations per minute (rpm).
* Temperature less than 95 degrees Fahrenheit (F) or 35 degrees Celsius (C).
* Tumor lysis syndrome.
* Sulfite allergy: amino acids administration are contraindicated. It is more common in steroid dependent asthmatics. (Please note that this is NOT sulfa allergy and is NOT contraindicated patients with sulfa allergy). Sulfites are present in dried fruits, beer, wines, sausages, jams, maple syrup, and many other food products.
* Serum sodium concentration < 130 mEq/L or > 150 mEq/L (Note: Once serum sodium levels are >= 130 or =< 150 mEq/L within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction.
* Serum creatinine level: Serum creatinine (SCr) > 2.5 mg/dL (Note: Once serum creatinine levels are =< 2.5 mg/dL within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction).
* Urine output < 400 cc/24 hours (hrs) plus creatinine > 2.5 mq/dl (Note: Once urine output levels are >= 400 cc within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction).
* Hyperkalemia K > 5.5 mEq/L (Note: Once potassium levels are =< 5.5 mEq/L within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction).
* Hyperglycemia: Glucose > 250 mg/dL (Note: Once glucose is below 250 mg/dL within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction.)
* Hyperphosphatemia: Serum phosphorous > 5.5 mg/dL.
* Patient with a history of metabolic abnormality in any one of the following amino acids: alanine, arginine, cysteine hydrochloride, glycine, histidine, isoleucine, leucine, lysine acetate, methionine, phenylalanine, phosphoric acid, proline, serine, threonine, tryptophan, and valine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L. Nates, MBA,MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 2019- December 2019
Groups:
- Intervention Group (EMR Solution): Standard of care + Early metabolic resuscitation
- Controlled Group (Standard Care): Received standard of care alone
Period: Overall Study
Arm/Group | Intervention Group (EMR Solution) | Controlled Group (Standard Care)
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the Intervention group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (EMR Solution) | Controlled Group (Standard Care) | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] |  | 52 [33 to 71] | 52 [33 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 2 | 2
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2
Cancer Type [Count of Participants; unit: Participants]
  Gastrointestinal | 0 | 0 | 0
  Breast | 0 | 0 | 0
  Lung | 0 | 1 | 1
Cancer stage [Count of Participants; unit: Participants]
  Metastatic Stage | 0 | 0 | 0
  Localized/Locally advanced | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 28-day Mortality
Description: To assess the efficacy of administering Early Metabolic Resuscitation with Standard of Care (SC + EMR) in patients diagnosed with septic shock for reducing 28-day mortality versus using the Standard of Care alone (SC). Twenty-eight day mortality is defined during the time from the day SC+EMR or SC was first administered until a patient dies or is followed through 28 days (whichever comes first).
Time Frame: up to 28 days or until death, whichever comes first
Population: No participants participated in the Intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (EMR Solution) | Controlled Group (Standard Care)
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With 90-Day Mortality
Description: To assess whether Early Metabolic Resuscitation with standard of care (SC + EMR) is an effective strategy to reduce ICU mortality, hospital mortality, and 90-day mortality of septic shock patients relative to SC. ICU mortality is defined as mortality at ICU discharge relative to SC.
Time Frame: up to 90 days or until death, whichever comes first
Population: No participants participated in the Intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (EMR Solution) | Controlled Group (Standard Care)
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Hospital Mortality
Description: To assess whether Early Metabolic Resuscitation with standard of care (SC + EMR) is an effective strategy to reduce hospital mortality of septic shock patients relative to SC.
Time Frame: up to 90 days or until death, whichever comes first
Population: No participants participated in the Intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (EMR Solution) | Controlled Group (Standard Care)
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With ICU Mortality
Description: To assess whether Early Metabolic Resuscitation with standard of care (SC + EMR) is an effective strategy to reduce ICU mortality of septic shock patients relative to SC. ICU mortality is defined as mortality at ICU discharge relative to SC.
Time Frame: up to 90-days or until death, whichever comes first
Population: No participants participated in the Intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (EMR Solution) | Controlled Group (Standard Care)
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline, up to 1 year
Description: No participants were enrolled in the Intervention Group
Arm/Group | Intervention Group (EMR Solution) | Controlled Group (Standard Care)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (EMR Solution) (N=0) | Controlled Group (Standard Care) (N=2)
Hypokalemia (Metabolism and nutrition disorders) | NA | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03895853/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03895853/ICF_001.pdf